CLINICAL TRIAL: NCT06176378
Title: A Clinical and Radiographic Evaluation of Low-Level Diode Laser Full Pulpotomy in Vital Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ehab Ali Elsayed, principal investigator/Assistant Lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 153/166
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Irreversible Pulpitis; Endodontic Inflammation
Keywords: Full pulpotomy; Low-level Diode Laser
MeSH Terms: conditions — Pulpitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Pulpotomy procedures (Experimental): In the traditional pulpotomy group, the coronal pulp was removed by the traditional method the the capping material applied
  Interventions: Other: traditional pulpotomy
- Diode laser Pulpotomy procedures (Experimental): in the low-level diode laser pulpotomy group, the radicular pulp was biostimulated using low-level diode laser before application of capping material
  Interventions: Device: diode laser pulpotomy

INTERVENTIONS:
Other: traditional pulpotomy — After complete deroofing, the coronal pulp was amputated to the level of the orifice using a high-speed size #2 round bur followed by rinsing the pulp chamber thoroughly with 5ml 0.9% saline solution.Hemostasis was then achieved by placing a sterile cotton pellet moistened with saline in the access cavity for 6 min.Retro MTA capping material was then applied,
  Other Names: full pulpotomy
  Arms: Traditional Pulpotomy procedures
Device: diode laser pulpotomy — after establishing hemostasis, low-level laser energy at (970nm, power .5W, duty cycle 50%, and frequency 5H) was applied to each pulp stump for 10 sec. through 320 microns optical fiber tip . The laser was used in pulsed non-contact mode at the level of the occlusal surface of the tooth.Retro MTA capping material was then applied,
  Other Names: laser biostimulation
  Arms: Diode laser Pulpotomy procedures

SUMMARY:
In this study, patients with symptoms of irreversible pulpitis in mature permanent molars were treated with two pulpotomies techniques after random allocation in either 2 groups: Diode laser pulpotomy and traditional pulpotomy using bioactive materials (retro mineral trioxide aggregate ) with each group.The null hypothesis of the study was there would be no difference in success rate between Diode laser and traditional methods of adult pulpotomy .

DETAILED DESCRIPTION:
In this study, 40 patients with symptoms of irreversible pulpitis in mature permanent 1st and 2nd molars were treated with two pulpotomy techniques after random allocation in either 2 groups: traditional pulpotomy and low-level diode laser pulpotomy. The pulp in each group was capped with Retro MTA . In the traditional pulpotomy group, the coronal pulp was removed by the traditional method while in the low-level diode laser pulpotomy group, the radicular pulp was biostimulated using low-level diode laser beam with parameters (970nm, power .5Watt, duty cycle 50%, and frequency 5H) 10 sec for each pulp stump in non-contact mode. After that, the capping material was prepared as manufacturer's instructions and applied over the pulp stamp, the final restoration was then placed in both groups. Patients were followed up after 6, 12, and 18 months to evaluate success and failure.

ELIGIBILITY:
Inclusion criteria:

* permanent 1st and 2nd molar
* irreversible pulpitis
* restorable

Exclusion criteria:

* Non-restorable teeth.
* Teeth with buccal restoration.
* Non-vital teeth that are not responsive to thermal stimuli or electric pulp test.
* Presence of swelling or sinus tracts.
* Teeth which showed sensitivity to percussion.
* Teeth with grade Ⅱ and Ⅲ mobility.
* Teeth with immature apices.
* Teeth with internal or external resorption or teeth with periapical pathosis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Assessment of success or failure | (T1): 1 week postoperative, (T2): after 6 months, (T3): after 12 months, and (T4) after 18 months.
  Assessment of success or failure was done using the technique described by Galeni et al
  Treatment was considered successful if the patient's final restoration was intact and the patient demonstrated no clinical symptoms (pain (spontaneous or on chewing), swelling, or sinus tract), and had a periapical index score of 1.
  • Treatment was considered uncertain if the patient's final restoration was intact, and the patient demonstrated no clinical symptoms (pain (spontaneous or on chewing), swelling, or sinus tract), and a PAI score of 2.
  •
  Treatment was considered a failure in the following situations:
  1. Any case in which the final restoration was not intact. Irrelevant clinical and radiographic symptoms.
  2. Any case in which the final restoration was intact and the patient demonstrated clinical symptoms. Irrelevant of PAI score.
  3. Any case in which the final restoration was intact and the patient had a PAI score of 3 or above. Irrelevant of clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt